CLINICAL TRIAL: NCT05185193
Title: Efficacy and Safety Evaluation of Changes in Lower Extremity Edema of Radiofrequency in Adult Women With Idiopathic Edema: Blinded, Cross-over, Pilot Study
Brief Title: Efficacy and Safety Evaluation of Changes in Lower Extremity Edema of Radiofrequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 03-2020-001
Record Dates: First submitted 2021-06-09; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Idiopathic Edema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency stimulation (Experimental): Participants received radiofrequency stimulation three times a day for 30 minutes once a day. After the end of the first session intervention, there was a washout period and the next intervention was started at a time point when the next menstruation was not likely (8-18 days after the onset of menstruation).
  Interventions: Device: radiofrequency
- sham stimulation (Sham Comparator): Participants received a sham stimulation similar to a radiofrequency stimulation three times a day for 30 minutes once a day. After the end of the first session intervention, there was a washout period and the next intervention was started at a time point when the next menstruation was not likely (8-18 days after the onset of menstruation).
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: radiofrequency — Radiofrequency of 9.50v, 218.5mA and 2.076W is applied once a day for 30 minutes, a total of 3 times
  Other Names: high frequency
  Arms: radiofrequency stimulation
Device: sham stimulation — The appearance is the same as the medical device for clinical trials, and when applied, the sound and the amount of light visible from the outside are designed to be the same as the medical device for clinical trials. The external light was the same, and only the high frequency that stimulates the dermis was blocked. The sham device was applied once a day for 30 minutes, a total of 3 times.
  Arms: sham stimulation

SUMMARY:
The purpose of this study is to verify the efficacy and safety of the radiofrequency stimulation compared to the sham stimulation in reducing lower extremity edema in adult women with idiopathic edema.

DETAILED DESCRIPTION:
In this study, based on the characteristics of radiofrequency, it was hypothesized that radiofrequency could have an effect on the reduction of lower extremity edema and prevention of fatigue. The occurrence of edema is interpreted as a problem that blood circulation is not smooth due to increased inflow of body fluid, and therefore the degree of edema is also used as an indicator of blood circulation.

Therefore, in this study, based on the principle that radiofrequency promotes phosphorylation and blood circulation, the purpose of this study is to investigate whether radiofrequency treatment is effective in reducing edema of the lower extremities and changing body heat in the lower extremities compared to the gastric stimulation device through exploratory research.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 19 and 72
2. Those who are not likely to menstruate during the trial treatment period (3 days) (females within 8 to 18 days after the onset of menstruation)
3. Those who meet the diagnostic criteria for idiopathic edema (McKendry criteria score of 15 or higher)
4. Those who show a weight change of 1.4 kg or more between morning and night measurements
5. Those who have a difference of 1cm or more from the ankle or 2cm or more from the calf when measuring the circumference in the morning and evening
6. Those who voluntarily agree to participate in this clinical trial and sign the consent form

Exclusion Criteria:

1. In the case of using a heart rate control device such as a metallic substance in the human body
2. During menstruation or if there is a possibility of pregnancy
3. If you have heart disease
4. If you have liver or kidney disease
5. If there is bleeding or internal bleeding from wounds or surgery
6. For hypertensive patients
7. For epilepsy patients
8. If you are taking weight loss or health-related drugs/health functional foods
9. In the case where it is judged by the principal investigator that participation in this study is not appropriate

Ages: 19 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Change of Circumference(the lower calf at 7 cm proximal to the midpoint of the medial malleolus, behind the medial malleolus, and the dorsum of the foot) | Changes of circumference before and immediately after 30 minutes radiofrequency stimulation on once a day basis in the experimental group
  Circumference was measured using a tape measure at three anatomical locations.

SECONDARY OUTCOMES:
Change of Volume | Changes of volume before and immediately after 30 minutes radiofrequency stimulation on once a day basis in the experimental group
  The leg volume test is measured using Volumeters (Deluxe Foot) of Jeongdo BNP Co., Ltd. in Korea.
  Measure using the principle of overflowing, fill a cylinder with a diameter of 30cm and a height of 30cm with water, put one leg in the cylinder with the ankle bent at 90 degrees, and take the overflowing water and measure the amount in ml.
digital infrared thermal imaging(DITI) | Changes of body heat before and immediately after 30 minutes radiofrequency stimulation on once a day basis in the experimental group
  Measure the subject's leg body heat using DITI.
Visual analog scale(VAS) | Changes of VAS score before and immediately after 30 minutes radiofrequency stimulation on once a day basis in the experimental group
  Discomfort VAS is used to measure the degree of discomfort for lower extremity edema after application of the device. And 0 indicates no discomfort at all, and 10 indicates the most severe discomfort imaginable.
weight | Changes of weight before and immediately after 30 minutes radiofrequency stimulation on once a day basis in the experimental group
  Measure the participant's weight (kg) using a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Il Shin, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan national university Yangsan Hospital, Gyeongsang, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No